CLINICAL TRIAL: NCT01411241
Title: Immunogenicity and Safety of a Booster Injection of DTaP-IPV//Hib (Pentaxim™) Administered Concomitantly With Tetravalent Dengue Vaccine in Healthy Toddlers Aged 15 to 18 Months in Mexico
Brief Title: Study of a Booster Injection of Pentaxim™ Vaccine Administered With Dengue Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYD33; U1111-1115-6290 (Other: WHO)
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Hemorrhagic Fever
Keywords: Dengue; Dengue Hemorrhagic Fever; CYD Dengue Vaccines; Pentaxim™
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Pentavac; Measles-Mumps-Rubella Vaccine; Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An observer-blind design was chosen since the products were visually different. For the second dose of CYD dengue vaccine, the person who administered the injections knew which product was administered while the subject/parent and Investigator were blinded. The first and third doses of CYD dengue vaccine were administered according to an open-label procedure. A placebo dose was administered at Month 7(Group 1) and concomitantly with Pentaxim vaccine at Month 6 (Group 2) to maintain the blind.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYD Dengue Vaccine Group 1 (Experimental): Participants received the first injection of CYD dengue vaccine at Month 0 (9 to 12 months of age), a measles, mumps, rubella (MMR) vaccine and pneumococcal conjugate vaccine at Month 1 (10 to 13 months of age), a booster dose of Pentaxim vaccine was administered concomitantly with the second injection of CYD dengue vaccine at Month 6 (15 to 18 months of age), placebo at Month 7 (16 to 19 months of age) to maintain the blind, and the third injection of CYD dengue vaccine at Month 12 (21 to 24 months).
  Interventions: Biological: Live, attenuated, recombinant dengue serotype 1, 2, 3, and 4 virus; Biological: DTaP IPV//Hib vaccine; Biological: Placebo; Biological: Measles, mumps, and rubella vaccine; Biological: Pneumococcal vaccine
- CYD Dengue Vaccine Group 2 (Experimental): Participants received the first injection of CYD dengue vaccine at Month 0 (9 to 12 months of age), a MMR vaccine and pneumococcal conjugate vaccine at Month 1 (10 to 13 months of age), the Pentaxim vaccine was administered concomitantly with placebo at Month 6 (15 to 18 months of age) to maintain the blind, a second injection of CYD dengue vaccine at Month 7 (16 to 19 months of age), and the third injection of CYD dengue vaccine at Month 12 (21 to 24 months).
  Interventions: Biological: Live, attenuated, recombinant dengue serotype 1, 2, 3, and 4 virus; Biological: DTaP IPV//Hib vaccine; Biological: Placebo; Biological: Measles, mumps, and rubella vaccine; Biological: Pneumococcal vaccine

INTERVENTIONS:
Biological: Live, attenuated, recombinant dengue serotype 1, 2, 3, and 4 virus — 0.5 mL, subcutaneous at age 9 to 12, 15 to 18 and 21 to 24 months.
  Other Names: CYD Dengue Vaccine
  Arms: CYD Dengue Vaccine Group 1
Biological: DTaP IPV//Hib vaccine — 0.5 mL, intramuscular
  Other Names: Pentaxim™
  Arms: CYD Dengue Vaccine Group 1
Biological: Placebo — 0.5 mL, subcutaneous
  Other Names: NaCl
  Arms: CYD Dengue Vaccine Group 1
Biological: Measles, mumps, and rubella vaccine — 0.5 mL, subcutaneous
  Other Names: Trimovax®
  Arms: CYD Dengue Vaccine Group 1
Biological: Pneumococcal vaccine — 0.5 mL, intramuscular
  Other Names: Prevenar®
  Arms: CYD Dengue Vaccine Group 1
Biological: Live, attenuated, recombinant dengue serotype 1, 2, 3, and 4 virus — 0.5 mL, subcutaneous at age 9 to 12, 16 to 19 and 21 to 24 months
  Other Names: CYD Dengue Vaccine
  Arms: CYD Dengue Vaccine Group 2
Biological: DTaP IPV//Hib vaccine — 0.5 mL, intramuscular
  Other Names: Pentaxim™
  Arms: CYD Dengue Vaccine Group 2
Biological: Placebo — 0.5 mL, subcutaneously
  Other Names: NaCl
  Arms: CYD Dengue Vaccine Group 2
Biological: Measles, mumps, and rubella vaccine — 0.5 mL, subcutaneous
  Other Names: Trimovax®
  Arms: CYD Dengue Vaccine Group 2
Biological: Pneumococcal vaccine — 0.5 mL, intramuscular
  Other Names: Prevenar®
  Arms: CYD Dengue Vaccine Group 2

SUMMARY:
The aim of the study was to assess whether the second CYD dengue vaccination could be administered concomitantly with the booster vaccination of a pediatric combination vaccine (Pentaxim™) during the same day visit but in 2 different sites of administration.

Primary Objective:

* To demonstrate the non-inferiority of the antibody response against all antigens (diphtheria, tetanus, pertussis, polio and Haemophilus influenzae type b (Hib)) in participants receiving one booster dose of Pentaxim™ vaccine administered concomitantly with the second dose of CYD dengue vaccine compared to participants receiving one booster dose of Pentaxim™ vaccine administered concomitantly with placebo.

Secondary Objectives:

* To describe the safety of Pentaxim™ vaccine administered concomitantly with the second dose of CYD dengue vaccine, or administered concomitantly with placebo.
* To describe the safety of the CYD dengue vaccine after the second dose of CYD dengue vaccine administered concomitantly with Pentaxim™ vaccine (at Visit 05) or administered alone (at Visit 06).
* To describe the safety of the CYD dengue vaccine in all participants after each dose.
* To describe the antibody response to each dengue virus serotype (post-Dose 2 and post-Dose 3) after the second dose of CYD dengue vaccine administered concomitantly with Pentaxim vaccine (at Visit 05) or administered alone (at Visit 06).
* To describe the antibody response to each dengue virus serotype post-Dose 2 and post-Dose 3.

DETAILED DESCRIPTION:
Participants required 8 or 9 clinic visits and received a total of 7 injections. The dengue post-vaccinal viremia was assessed at Visit 2 from a subset of toddlers. The dengue immunogenicity was assessed 28 days after CYD dengue dose 2 and dose 3 from a subset of toddlers. Participants were followed-up for safety after each vaccine dose and for 6 months after the last dengue vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 to 12 months on the day of inclusion.
* Born at full term of pregnancy (>= 37 weeks) and with a birth weight >= 2.5 kg.
* Participant in good health, based on medical history and physical examination.
* Documentation of completion of the primary vaccination series with Pentaxim vaccine with the 3 doses received between 2 and 8 months of age.
* Informed consent form had been signed and dated by both parents or other legally acceptable representative (and by 2 mandatory witnesses as required by local regulations).
* Participant and parent/guardian attended all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination.
* Previous vaccination against flavivirus diseases, measles, mumps, rubella, previous booster vaccination against pneumococcal diseases, diphtheria, tetanus, pertussis, Hib and/or polio.
* Receipt of blood or blood-derived products in the past 3 months which might interfere with assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Personal seropositivity for human immunodeficiency virus (HIV) or hepatitis C as reported by the parent(s)/legally acceptable representative.
* History of pertussis and/or Hib infection as reported by the parent(s)/legally acceptable representative.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* History of contraindication to the receipt of vaccines containing components of Pentaxim vaccine (diphtheria toxoid, tetanus toxoid, pertussis toxoid, filamentous hemagglutinin, polyribosylribitol phosphate [PRP] and polio) or of measles, mumps and rubella vaccine and of pneumococcal vaccine.
* Thrombocytopenia, as reported by the parent(s)/legally acceptable representative.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* History of central nervous system disorder or disease, including seizures.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Identified as a child (adopted or natural) of the Investigator or of site employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center.

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2011-07-18 (Actual); Primary Completion 2014-02-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (4):
- Mexico (4):
  - Acapulco de Juárez, Guerrero
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Mérida, Yucatán

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 18 July 2011 to 31 July 2012 at 3 clinical sites in Mexico. The study planned for 732 participants; however, recruitment was stopped when 720 participants were enrolled due to the difficulty in enrolling participants.
Pre-assignment Details: A total of 720 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled, out of which 309 participants were randomized to Group 1 and 315 in Group 2, and 96 participants were not randomized to Group 1 or 2.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Started | 309 | 315
Completed | 298 | 293
Not Completed | 11 | 22
Not completed — Protocol Violation | 0 | 5
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Serious Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- CYD Dengue Vaccine Group 1: Participants received the first injection of CYD dengue vaccine at Month 0 (9 to 12 months of age), a MMR vaccine and pneumococcal conjugate vaccine at Month 1 (10 to 13 months of age), a booster dose of Pentaxim vaccine was administered concomitantly with the second injection of CYD dengue vaccine at Month 6 (15 to 18 months of age), placebo at Month 7 (16 to 19 months of age) to maintain the blind, and the third injection of CYD dengue vaccine at Month 12 (21 to 24 months).
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2 | Total
Number analyzed (Participants) | 309 | 315 | 624
Age, Customized [Count of Participants; unit: Participants]
  1 month to 23 months | 309 | 315 | 624
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 139 | 285
  Male | 163 | 176 | 339

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroprotection or Booster Response After a Booster Injection (Inj.) of Diphtheria, Tetanus, Acellular Pertussis(DTaP)-Inactivated Polio Virus (IPV)//Hib (Pentaxim™) Administered Concomitantly With CYD Dengue Vaccine
Description: Antibodies (Ab) against diphtheria, tetanus toxoid, pertussis toxoid (PT), and filamentous hemaglutinin (FHA) was measured by enzyme-linked immunosorbent assay (ELISA), polyribosylribitol phosphate (PRP) by Farr-type radioimmunoassay, and poliovirus types 1, 2, and 3 by seroneutralization assay. Seroprotection was defined as >=0.1 International Unit (IU)/mL for diphtheria toxoid and tetanus toxoid, >=8 1/dil for poliovirus types 1, 2, and 3, and >=1.0 μg/mL for PRP. Booster response to PT and FHA: participants whose pre-vaccination Ab titers were < lower limit of quantitation (LLOQ), a booster response occurred if they had post-vaccination levels >=4* LLOQ; participants whose pre-vaccination Ab concentrations were >=LLOQ but <4* LLOQ, a booster response occurred if they had a 4-fold increase (post/pre-vaccination levels >=4); for participants whose pre-vaccination Ab concentrations were >=4* LLOQ, a booster response occurred if they had a 2-fold increase (post/pre-vaccination >=2).
Time Frame: 28 days post-injection
Population: Per-protocol analysis set:all participants who had no protocol deviations (not meet inclusion/exclusion criteria,not received vaccine in time window, administration not done per protocol) and could impact Pentaxim vaccine immunogenicity up to Visit 06 (Month 07). Here, 'number analyzed'=participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 256 | 270
Percentage of participants
  Anti-diphtheria: number analyzed (Participants) | 255 | 270
  Anti-diphtheria | 100.0 | 100.0
  Anti-tetanus: number analyzed (Participants) | 255 | 270
  Anti-tetanus | 100.0 | 99.6
  Anti-polio 1: number analyzed (Participants) | 256 | 269
  Anti-polio 1 | 100.0 | 99.6
  Anti-polio 2 | 100.0 | 100.0
  Anti-polio 3: number analyzed (Participants) | 254 | 267
  Anti-polio 3 | 100 | 99.6
  Anti-PRP | 100.0 | 100.0
  Anti-PT: number analyzed (Participants) | 255 | 269
  Anti-PT | 96.5 | 97.0
  Anti-FHA | 93.0 | 93.3
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group 1 vs CYD Dengue Vaccine Group 2; Non-inferiority (Group 1 - Group 2); Anti-diphtheria. Non-inferiority of Pentaxim booster dose based on seroprotection/booster response was assessed 28 days after injection; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of all the 95% Confidence Interval (CI) of the difference is greater than -10% for all antigens. Wilson score (without continuity adjustment) 95% two-sided CI was used for the difference of seroprotection/booster rates; Difference in percentage = 0.0, 95% CI 2-sided [-1.48 to 1.40]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Group 1 vs CYD Dengue Vaccine Group 2; Non-inferiority (Group 1 - Group 2); Anti-tetanus. Non-inferiority of Pentaxim booster dose based on seroprotection/booster response was assessed 28 days after injection; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of all the 95% CI of the difference is greater than -10% for all antigens. Wilson score (without continuity adjustment) 95% two-sided CI was used for the difference of seroprotection/booster rates; Difference in percentage = 0.37, 95% CI 2-sided [-1.14 to 2.07]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Group 1 vs CYD Dengue Vaccine Group 2; Non-inferiority (Group 1 - Group 2); Anti-polio 1. Non-inferiority of Pentaxim booster dose based on seroprotection/booster response was assessed 28 days after injection; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = 0.37, 95% CI 2-sided [-1.14 to 2.08]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Group 1 vs CYD Dengue Vaccine Group 2; Non-inferiority (Group 1 - Group 2); Anti-polio 2. Non-inferiority of Pentaxim booster dose based on seroprotection/booster response was assessed 28 days after injection; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = 0.0, 95% CI 2-sided [-1.48 to 1.40]
Statistical Analysis 5: Comparison: CYD Dengue Vaccine Group 1 vs CYD Dengue Vaccine Group 2; Non-inferiority (Group 1 - Group 2); Anti-polio 3. Non-inferiority of Pentaxim booster dose based on seroprotection/booster response was assessed 28 days after injection; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = 0.37, 95% CI 2-sided [-1.15 to 2.09]
Statistical Analysis 6: Comparison: CYD Dengue Vaccine Group 1 vs CYD Dengue Vaccine Group 2; Non-inferiority (Group 1 - Group 2); Anti-PRP. Non-inferiority of Pentaxim booster dose based on seroprotection/booster response was assessed 28 days after injection; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = 0.0, 95% CI 2-sided [-1.48 to 1.40]
Statistical Analysis 7: Comparison: CYD Dengue Vaccine Group 1 vs CYD Dengue Vaccine Group 2; Non-inferiority (Group 1 - Group 2); Anti-PT. Non-inferiority of Pentaxim booster dose based on seroprotection/booster response was assessed 28 days after injection; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = -0.56, 95% CI 2-sided [-3.93 to 2.69]
Statistical Analysis 8: Comparison: CYD Dengue Vaccine Group 1 vs CYD Dengue Vaccine Group 2; Non-inferiority (Group 1 - Group 2); Anti-FHA. Non-inferiority of Pentaxim booster dose based on seroprotection/booster response was assessed 28 days after injection; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = -0.36, 95% CI 2-sided [-4.87 to 4.06]

2. Secondary Outcome: Geometric Mean Titers Against Each Serotype With the Parental Dengue Virus Strains Before and After a Booster Injection of DTaP-IPV//Hib (Pentaxim™) Administered Concomitantly With CYD Dengue Vaccine
Description: Geometric mean titers of antibodies against the dengue virus serotypes were measured by dengue plaque reduction neutralization test (PRNT).
Time Frame: Pre-injection 1 and 28 days post-injection 2 and 3
Population: Analysis was performed on Full analysis set for dengue immunogenicity which included participants randomized into the dengue immunogenicity subset who received at least one dose of CYD dengue vaccine. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 109 | 107
Titers (1/dilution)
  Serotype 1; Pre-injection 1 | 5.28 [4.82 to 5.78] | 5.35 [4.85 to 5.91]
  Serotype 1; Post-injection 2: number analyzed (Participants) | 105 | 103
  Serotype 1; Post-injection 2 | 39.8 [30.5 to 51.9] | 62.8 [48.1 to 82.0]
  Serotype 1; Post-injection 3: number analyzed (Participants) | 102 | 98
  Serotype 1; Post-injection 3 | 93.1 [76.6 to 113] | 97.0 [78.8 to 120]
  Serotype 2; Pre-injection 1 | 5.22 [4.89 to 5.57] | 5.53 [5.04 to 6.07]
  Serotype 2; Post-injection 2: number analyzed (Participants) | 105 | 103
  Serotype 2; Post-injection 2 | 109 [80.2 to 149] | 121 [89.3 to 164]
  Serotype 2; Post-injection 3: number analyzed (Participants) | 102 | 98
  Serotype 2; Post-injection 3 | 189 [156 to 228] | 208 [166 to 261]
  Serotype 3; Pre-injection 1 | 5.26 [4.93 to 5.62] | 5.38 [4.95 to 5.84]
  Serotype 3; Post-injection 2: number analyzed (Participants) | 105 | 103
  Serotype 3; Post-injection 2 | 92.8 [75.7 to 114] | 116 [91.1 to 149]
  Serotype 3; Post-injection 3: number analyzed (Participants) | 102 | 98
  Serotype 3; Post-injection 3 | 196 [168 to 229] | 217 [183 to 256]
  Serotype 4; Pre-injection 1: number analyzed (Participants) | 109 | 106
  Serotype 4; Pre-injection 1 | 5.11 [4.94 to 5.28] | 5.00 [5.00 to 5.00]
  Serotype 4; Post-injection 2: number analyzed (Participants) | 105 | 103
  Serotype 4; Post-injection 2 | 57.8 [44.5 to 75.2] | 104 [81.7 to 131]
  Serotype 4; Post-injection 3: number analyzed (Participants) | 102 | 98
  Serotype 4; Post-injection 3 | 121 [103 to 142] | 127 [103 to 155]

3. Secondary Outcome: Geometric Mean Titer Ratios Against Each Serotype With the Parental of Dengue Virus Strains Before and After a Booster Injection of DTaP-IPV//Hib (Pentaxim™) Administered Concomitantly With CYD Dengue Vaccine
Description: Geometric mean titers of antibodies against the dengue virus serotypes were measured by dengue PRNT.
Time Frame: Pre-injection 1 and 28 days post-injection 2 and 3
Population: Analysis was performed on Full analysis set for dengue immunogenicity. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 109 | 107
Titer ratio
  Serotype 1: Post-inj 2 value/pre-inj 1 value: number analyzed (Participants) | 105 | 103
  Serotype 1: Post-inj 2 value/pre-inj 1 value | 3.81 [2.95 to 4.93] | 5.97 [4.64 to 7.68]
  Serotype 1: Post-inj 3 value/pre-inj 1 value: number analyzed (Participants) | 102 | 98
  Serotype 1: Post-inj 3 value/pre-inj 1 value | 8.91 [7.40 to 10.7] | 9.20 [7.55 to 11.2]
  Serotype 2: Post-inj 2 value/pre-inj 1 value: number analyzed (Participants) | 105 | 103
  Serotype 2: Post-inj 2 value/pre-inj 1 value | 10.6 [7.77 to 14.5] | 11.5 [8.50 to 15.4]
  Serotype 2: Post-inj 3 value/pre-inj 1 value: number analyzed (Participants) | 102 | 98
  Serotype 2: Post-inj 3 value/pre-inj 1 value | 18.3 [15.1 to 22.1] | 19.6 [15.6 to 24.7]
  Serotype 3: Post-inj 2 value/pre-inj 1 value: number analyzed (Participants) | 105 | 103
  Serotype 3: Post-inj 2 value/pre-inj 1 value | 8.97 [7.33 to 11.0] | 11.1 [8.73 to 14.1]
  Serotype 3: Post-inj 3 value/pre-inj 1 value: number analyzed (Participants) | 102 | 98
  Serotype 3: Post-inj 3 value/pre-inj 1 value | 19.1 [16.4 to 22.2] | 20.6 [17.4 to 24.4]
  Serotype 4: Post-inj 2 value/pre-inj 1 value: number analyzed (Participants) | 105 | 102
  Serotype 4: Post-inj 2 value/pre-inj 1 value | 5.73 [4.40 to 7.45] | 10.0 [7.96 to 12.6]
  Serotype 4: Post-inj 3 value/pre-inj 1 value: number analyzed (Participants) | 102 | 97
  Serotype 4: Post-inj 3 value/pre-inj 1 value | 12.0 [10.2 to 14.1] | 12.6 [10.3 to 15.5]

4. Secondary Outcome: Percentage of Participants With a Seropositivity Against Each Serotype With the Parental Dengue Virus Strains Before and After a Booster Injection of DTaP-IPV//Hib (Pentaxim™) Administered Concomitantly With CYD Dengue Vaccine
Description: Seropositivity against each dengue virus serotype (parental strains) were measured by dengue PRNT. Seropositivity was defined as antibody titers >=10 (1/dilution).
Time Frame: Pre-injection 1 and 28 days post-injection 2 and 3
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 109 | 107
Percentage of participants
  Serotype 1; Pre-injection 1 | 1.8 | 2.8
  Serotype 1; Post-injection 2: number analyzed (Participants) | 105 | 103
  Serotype 1; Post-injection 2 | 84.8 | 92.2
  Serotype 1; Post-injection 3: number analyzed (Participants) | 102 | 98
  Serotype 1; Post-injection 3 | 100.0 | 100.0
  Serotype 2; Pre-injection 1 | 1.8 | 4.7
  Serotype 2; Post-injection 2: number analyzed (Participants) | 105 | 103
  Serotype 2; Post-injection 2 | 98.1 | 96.1
  Serotype 2; Post-injection 3: number analyzed (Participants) | 102 | 98
  Serotype 2; Post-injection 3 | 100.0 | 100.0
  Serotype 3; Pre-injection 1 | 2.8 | 3.7
  Serotype 3; Post-injection 2: number analyzed (Participants) | 105 | 103
  Serotype 3; Post-injection 2 | 100.0 | 98.1
  Serotype 3; Post-injection 3: number analyzed (Participants) | 102 | 98
  Serotype 3; Post-injection 3 | 100.0 | 100.0
  Serotype 4; Pre-injection 1: number analyzed (Participants) | 109 | 106
  Serotype 4; Pre-injection 1 | 1.8 | 0.0
  Serotype 4; Post-injection 2: number analyzed (Participants) | 105 | 103
  Serotype 4; Post-injection 2 | 90.5 | 96.1
  Serotype 4; Post-injection 3: number analyzed (Participants) | 102 | 98
  Serotype 4; Post-injection 3 | 100.0 | 100.0

5. Secondary Outcome: Percentage of Participants With Seropositivity Against at Least One, Two, Three, or Four Serotypes With the Parental Dengue Virus Strains Before and After a Booster Injection of DTaP-IPV// Hib (Pentaxim™) Administered With CYD Dengue Vaccine
Description: as for outcome 4
Time Frame: Pre-injection 1 and 28 days post-injection 2 and 3
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 109 | 107
Percentage of participants
  At least 1 serotype; Pre-injection 1 | 4.6 | 8.4
  At least 1 serotype; Post-injection 2: number analyzed (Participants) | 105 | 103
  At least 1 serotype; Post-injection 2 | 100.0 | 100.0
  At least 1 serotype; Post-injection 3: number analyzed (Participants) | 102 | 98
  At least 1 serotype; Post-injection 3 | 100.0 | 100.0
  At least 2 serotypes; Pre-injection 1 | 1.8 | 1.9
  At least 2 serotypes; Post-injection 2: number analyzed (Participants) | 105 | 103
  At least 2 serotypes; Post-injection 2 | 100.0 | 98.1
  At least 2 serotypes; Post-injection 3: number analyzed (Participants) | 102 | 98
  At least 2 serotypes; Post-injection 3 | 100.0 | 100.0
  At least 3 serotypes; Pre-injection 1 | 0.9 | 0.9
  At least 3 serotypes; Post-injection 2: number analyzed (Participants) | 105 | 103
  At least 3 serotypes; Post-injection 2 | 94.3 | 95.1
  At least 3 serotypes; Post-injection 3: number analyzed (Participants) | 102 | 98
  At least 3 serotypes; Post-injection 3 | 100.0 | 100.0
  All 4 serotypes; Pre-injection 1 | 0.9 | 0.0
  All 4 serotypes; Post-injection 2: number analyzed (Participants) | 105 | 103
  All 4 serotypes; Post-injection 2 | 79.0 | 89.3
  All 4 serotypes; Post-injection 3: number analyzed (Participants) | 102 | 98
  All 4 serotypes; Post-injection 3 | 100.0 | 100.0

6. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site and Systemic Reactions Following the First Injection With CYD Dengue Vaccine
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling. Solicited systemic reactions: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability. Grade (Grd) 3 Solicited injection site reactions: Tenderness, cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling: >=50 mm. Grade 3 Solicited systemic reactions: Fever: >39.5 degree Celsius (°C); Vomiting: >=6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal: >3 hours; Drowsiness: Sleeping most of the time or difficult to wake up; Appetite lost: refuses >=3 feeds/meals or refuses most feeds/meals; Irritability: inconsolable.
Time Frame: Day 0 up to Day 14 post-first injection
Population: Analysis was performed on Safety analysis set which included participants who received at least one dose of CYD dengue vaccine, Pentaxim vaccine or placebo. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 309 | 315
Percentage of participants
  Injection site Tenderness: number analyzed (Participants) | 308 | 312
  Injection site Tenderness | 29.9 | 33.3
  Grade 3 Injection site Tenderness: number analyzed (Participants) | 308 | 312
  Grade 3 Injection site Tenderness | 0.3 | 0.0
  Injection site Erythema: number analyzed (Participants) | 308 | 312
  Injection site Erythema | 14.0 | 15.7
  Grade 3 Injection site Erythema: number analyzed (Participants) | 308 | 312
  Grade 3 Injection site Erythema | 0.0 | 0.0
  Injection site Swelling: number analyzed (Participants) | 308 | 312
  Injection site Swelling | 4.9 | 10.9
  Grade 3 Injection site Swelling: number analyzed (Participants) | 308 | 312
  Grade 3 Injection site Swelling | 0.0 | 0.3
  Fever: number analyzed (Participants) | 307 | 313
  Fever | 25.1 | 28.1
  Grade 3 Fever: number analyzed (Participants) | 307 | 313
  Grade 3 Fever | 1.6 | 0.0
  Vomiting: number analyzed (Participants) | 308 | 312
  Vomiting | 18.8 | 17.6
  Grade 3 Vomiting: number analyzed (Participants) | 308 | 312
  Grade 3 Vomiting | 1.3 | 0.6
  Crying abnormal: number analyzed (Participants) | 308 | 312
  Crying abnormal | 36.4 | 38.5
  Grade 3 Crying abnormal: number analyzed (Participants) | 308 | 312
  Grade 3 Crying abnormal | 2.3 | 2.2
  Drowsiness: number analyzed (Participants) | 308 | 312
  Drowsiness | 24.0 | 23.4
  Grade 3 Drowsiness: number analyzed (Participants) | 308 | 312
  Grade 3 Drowsiness | 1.9 | 1.6
  Appetite lost: number analyzed (Participants) | 308 | 311
  Appetite lost | 32.5 | 34.7
  Grade 3 Appetite lost: number analyzed (Participants) | 308 | 311
  Grade 3 Appetite lost | 4.5 | 4.5
  Injection site Irritability: number analyzed (Participants) | 308 | 312
  Injection site Irritability | 47.1 | 45.5
  Grade 3 Injection site Irritability: number analyzed (Participants) | 308 | 312
  Grade 3 Injection site Irritability | 3.2 | 4.2

7. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site and Systemic Reactions Following a Booster Injection of DTaP-IPV// Hib (Pentaxim™) Administered Concomitantly With Either CYD Dengue Vaccine or a Placebo Vaccine
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling. Solicited systemic reactions: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability. Grade 3 Solicited injection site reactions: Tenderness: cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling: >=50 mm. Grade 3 Solicited systemic reactions: Fever: >39.5°C; Vomiting: >=6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal: >3 hours; Drowsiness: sleeping most of the time or difficult to wake up; Appetite lost: refuses >=3 feeds/meals or refuses most feeds/meals; Irritability: inconsolable; and Extensive swelling, severe.
Time Frame: Day 0 up to Day 14 post-booster injection
Population: Analysis was performed on Safety analysis set. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 309 | 314
Percentage of participants
  Injection site Tenderness: number analyzed (Participants) | 301 | 305
  Injection site Tenderness | 43.2 | 42.3
  Grade 3 Injection site Tenderness: number analyzed (Participants) | 301 | 305
  Grade 3 Injection site Tenderness | 1.0 | 0.7
  Injection site Tenderness; Post- Pentaxim: number analyzed (Participants) | 301 | 305
  Injection site Tenderness; Post- Pentaxim | 37.5 | 37.7
  Grade 3 Injection site Tenderness; Post- Pentaxim: number analyzed (Participants) | 301 | 305
  Grade 3 Injection site Tenderness; Post- Pentaxim | 1.0 | 0.7
  Injection site Tenderness; Post-CYD dengue/placebo: number analyzed (Participants) | 301 | 305
  Injection site Tenderness; Post-CYD dengue/placebo | 33.2 | 30.5
  Grd 3 Inj. site Tenderness;Post-CYD dengue/placebo: number analyzed (Participants) | 301 | 305
  Grd 3 Inj. site Tenderness;Post-CYD dengue/placebo | 0.0 | 0.3
  Injection site Erythema: number analyzed (Participants) | 301 | 305
  Injection site Erythema | 15.0 | 20.3
  Grade 3 Injection site Erythema: number analyzed (Participants) | 301 | 305
  Grade 3 Injection site Erythema | 0.3 | 0.0
  Injection site Erythema; Post-Pentaxim: number analyzed (Participants) | 301 | 304
  Injection site Erythema; Post-Pentaxim | 13.0 | 17.8
  Grade 3 Injection site Erythema; Post- Pentaxim: number analyzed (Participants) | 301 | 304
  Grade 3 Injection site Erythema; Post- Pentaxim | 0.3 | 0.0
  Injection site Erythema; Post-CYD dengue/placebo: number analyzed (Participants) | 301 | 305
  Injection site Erythema; Post-CYD dengue/placebo | 8.3 | 13.1
  Grd 3 Inj. site Erythema; Post-CYD dengue/placebo: number analyzed (Participants) | 301 | 305
  Grd 3 Inj. site Erythema; Post-CYD dengue/placebo | 0.0 | 0.0
  Injection site Swelling: number analyzed (Participants) | 301 | 305
  Injection site Swelling | 11.6 | 17.0
  Grade 3 Injection site Swelling: number analyzed (Participants) | 301 | 305
  Grade 3 Injection site Swelling | 0.3 | 0.0
  Injection site Swelling; Post-Pentaxim: number analyzed (Participants) | 299 | 305
  Injection site Swelling; Post-Pentaxim | 9.4 | 16.1
  Grade 3 Injection site Swelling; Post- Pentaxim: number analyzed (Participants) | 299 | 305
  Grade 3 Injection site Swelling; Post- Pentaxim | 0.3 | 0.0
  Injection site Swelling; Post-CYD dengue/placebo: number analyzed (Participants) | 301 | 305
  Injection site Swelling; Post-CYD dengue/placebo | 5.0 | 7.2
  Grd 3 Inj. site Swelling; Post-CYD dengue/placebo: number analyzed (Participants) | 301 | 305
  Grd 3 Inj. site Swelling; Post-CYD dengue/placebo | 0.0 | 0.0
  Injection site extensive swelling; Post- Pentaxim: number analyzed (Participants) | 301 | 306
  Injection site extensive swelling; Post- Pentaxim | 0.0 | 0.0
  Grd 3 Inj. site extensive swelling; Post- Pentaxim: number analyzed (Participants) | 301 | 306
  Grd 3 Inj. site extensive swelling; Post- Pentaxim | 0.0 | 0.0
  Fever: number analyzed (Participants) | 299 | 300
  Fever | 29.1 | 24.3
  Grade 3 Fever: number analyzed (Participants) | 299 | 300
  Grade 3 Fever | 1.0 | 0.0
  Vomiting: number analyzed (Participants) | 300 | 305
  Vomiting | 11.7 | 11.8
  Grade 3 Vomiting: number analyzed (Participants) | 300 | 305
  Grade 3 Vomiting | 1.0 | 0.0
  Crying abnormal: number analyzed (Participants) | 300 | 305
  Crying abnormal | 33.7 | 30.8
  Grade 3 Crying abnormal: number analyzed (Participants) | 300 | 305
  Grade 3 Crying abnormal | 0.7 | 1.6
  Drowsiness: number analyzed (Participants) | 300 | 305
  Drowsiness | 19.7 | 17.0
  Grade 3 Drowsiness: number analyzed (Participants) | 300 | 305
  Grade 3 Drowsiness | 1.0 | 0.7
  Appetite lost: number analyzed (Participants) | 300 | 305
  Appetite lost | 23.3 | 23.0
  Grade 3 Appetite lost: number analyzed (Participants) | 300 | 305
  Grade 3 Appetite lost | 3.7 | 3.0
  Irritability: number analyzed (Participants) | 300 | 305
  Irritability | 37.7 | 39.7
  Grade 3 Irritability: number analyzed (Participants) | 300 | 305
  Grade 3 Irritability | 1.0 | 0.7

8. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site and Systemic Reactions Following a Second Injection of CYD Dengue Vaccine or a Placebo Vaccine
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling. Solicited systemic reactions: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability. Grade 3 Solicited injection site reactions: Tenderness: cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling: >=50 mm. Grade 3 Solicited systemic reactions: Fever: >39.5°C; Vomiting: >=6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal: >3 hours; Drowsiness, Sleeping most of the time or difficult to wake up; Appetite lost: refuses >=3 feeds/meals or refuses most feeds/meals; Irritability: inconsolable.
Time Frame: Day 0 up to Day 14 post-second injection
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 301 | 302
Percentage of participants
  Injection site Tenderness: number analyzed (Participants) | 294 | 296
  Injection site Tenderness | 24.5 | 25.7
  Grade 3 Injection site Tenderness: number analyzed (Participants) | 294 | 296
  Grade 3 Injection site Tenderness | 0.0 | 0.0
  Injection site Erythema: number analyzed (Participants) | 294 | 296
  Injection site Erythema | 8.2 | 10.1
  Grade 3 Injection site Erythema: number analyzed (Participants) | 294 | 296
  Grade 3 Injection site Erythema | 0.0 | 0.0
  Injection site Swelling: number analyzed (Participants) | 294 | 296
  Injection site Swelling | 4.4 | 5.1
  Grade 3 Injection site Swelling: number analyzed (Participants) | 294 | 296
  Grade 3 Injection site Swelling | 0.0 | 0.3
  Fever: number analyzed (Participants) | 293 | 293
  Fever | 16.7 | 18.1
  Grade 3 Fever: number analyzed (Participants) | 293 | 293
  Grade 3 Fever | 0.0 | 0.7
  Vomiting: number analyzed (Participants) | 293 | 296
  Vomiting | 6.8 | 8.8
  Grade 3 Vomiting: number analyzed (Participants) | 293 | 296
  Grade 3 Vomiting | 0.3 | 0.0
  Crying abnormal: number analyzed (Participants) | 293 | 296
  Crying abnormal | 21.2 | 24.3
  Grade 3 Crying abnormal: number analyzed (Participants) | 293 | 296
  Grade 3 Crying abnormal | 0.0 | 0.3
  Drowsiness: number analyzed (Participants) | 293 | 296
  Drowsiness | 11.9 | 14.9
  Grade 3 Drowsiness: number analyzed (Participants) | 293 | 296
  Grade 3 Drowsiness | 0.0 | 0.0
  Appetite lost: number analyzed (Participants) | 293 | 296
  Appetite lost | 17.7 | 20.9
  Grade 3 Appetite lost: number analyzed (Participants) | 293 | 296
  Grade 3 Appetite lost | 1.7 | 1.7
  Irritability: number analyzed (Participants) | 293 | 296
  Irritability | 23.9 | 25.3
  Grade 3 Irritability: number analyzed (Participants) | 293 | 296
  Grade 3 Irritability | 0.3 | 1.0

9. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site and Systemic Reactions Following a Third Injection of CYD Dengue Vaccine
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling. Solicited systemic reactions: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability. Grade 3 Solicited injection site reactions: Tenderness: cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling: >=50 mm. Grade 3 Solicited systemic reactions: Fever: >39.5°C; Vomiting: >=6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal: >3 hours; Drowsiness: sleeping most of the time or difficult to wake up; Appetite lost: refuses >=3 feeds/meals or refuses most feeds/meals; Irritability: inconsolable.
Time Frame: Day 0 up to Day 14 post-third injection
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
Number analyzed (Participants) | 298 | 297
Percentage of participants
  Injection site Tenderness: number analyzed (Participants) | 298 | 291
  Injection site Tenderness | 19.8 | 25.4
  Grade 3 Injection site Tenderness: number analyzed (Participants) | 298 | 291
  Grade 3 Injection site Tenderness | 0.0 | 0.0
  Injection site Erythema: number analyzed (Participants) | 298 | 291
  Injection site Erythema | 6.7 | 5.8
  Grade 3 Injection site Erythema: number analyzed (Participants) | 298 | 291
  Grade 3 Injection site Erythema | 0.0 | 0.0
  Injection site Swelling: number analyzed (Participants) | 298 | 291
  Injection site Swelling | 2.0 | 2.7
  Grade 3 Injection site Swelling: number analyzed (Participants) | 298 | 291
  Grade 3 Injection site Swelling | 0.0 | 0.0
  Fever: number analyzed (Participants) | 294 | 289
  Fever | 16.0 | 15.2
  Grade 3 Fever: number analyzed (Participants) | 294 | 289
  Grade 3 Fever | 1.0 | 0.0
  Vomiting: number analyzed (Participants) | 298 | 291
  Vomiting | 4.4 | 7.2
  Grade 3 Vomiting: number analyzed (Participants) | 298 | 291
  Grade 3 Vomiting | 0.7 | 1.0
  Crying abnormal: number analyzed (Participants) | 298 | 291
  Crying abnormal | 21.5 | 18.9
  Grade 3 Crying abnormal: number analyzed (Participants) | 298 | 291
  Grade 3 Crying abnormal | 0.7 | 0.3
  Drowsiness: number analyzed (Participants) | 298 | 291
  Drowsiness | 10.4 | 10.0
  Grade 3 Drowsiness: number analyzed (Participants) | 298 | 291
  Grade 3 Drowsiness | 0.7 | 0.7
  Appetite lost: number analyzed (Participants) | 298 | 291
  Appetite lost | 18.8 | 18.6
  Grade 3 Appetite lost: number analyzed (Participants) | 298 | 291
  Grade 3 Appetite lost | 1.3 | 2.4
  Irritability: number analyzed (Participants) | 298 | 291
  Irritability | 23.8 | 20.6
  Grade 3 Irritability: number analyzed (Participants) | 298 | 291
  Grade 3 Irritability | 1.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to 6 months post-third CYD injection (up to 18 months).
Description: Analysis was performed on Safety analysis set.
Arm/Group | CYD Dengue Vaccine Group 1 | CYD Dengue Vaccine Group 2
All-Cause Mortality (participants affected / at risk) | 0/309 | 1/315
Serious Adverse Events (participants affected / at risk) | 17/309 | 21/315
Other Adverse Events (participants affected / at risk) | 145/309 | 142/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group 1 (N=309) | CYD Dengue Vaccine Group 2 (N=315)
Accidental exposure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 5 (6) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0)
Ascariasis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 2 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYD Dengue Vaccine Group 1 (N=309) | CYD Dengue Vaccine Group 2 (N=315)
Drowsiness; Post-injection 1 (Nervous system disorders) | 74/308 (74) | 73/312 (73)
Injection site Tenderness; Post-injection 1 (General disorders) | 92 (92) | 104/312 (104)
Injection site Erythema; Post-injection 1 (General disorders) | 43/308 (43) | 49/312 (49)
Injection site Swelling; Post-injection 1 (General disorders) | 15/308 (15) | 34/312 (34)
Fever; Post-injection 1 (General disorders) | 77/307 (77) | 88/313 (88)
Crying abnormal; Post-injection 1 (Psychiatric disorders) | 112/308 (112) | 120/312 (120)
Irritability; Post-injection 1 (Psychiatric disorders) | 145/308 (145) | 142/312 (142)
Diarrhoea (Gastrointestinal disorders) | 34 (41) | 34 (37)
Vomiting; Post-injection 1 (Gastrointestinal disorders) | 58/308 (58) | 55/312 (55)
Appetite lost; Post-injection 1 (Metabolism and nutrition disorders) | 100/308 (100) | 108/311 (108)
Gastroenteritis (Infections and infestations) | 55 (61) | 47 (51)
Nasopharyngitis (Infections and infestations) | 109 (147) | 104 (132)
Pharyngitis (Infections and infestations) | 50 (60) | 57 (69)
Pharyngotonsillitis (Infections and infestations) | 24 (28) | 33 (33)
Rhinitis (Infections and infestations) | 25 (26) | 22 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.